CLINICAL TRIAL: NCT04655703
Title: A Phase 4, Prospective, Randomized Trial to Evaluate Postoperative Outcomes in Total Knee Arthroplasy Patients Using the DJO X4 Brace With the Motion Intelligence Platform
Brief Title: Use of the DJO Brace With the Motion Intelligence Platform in the Postoperative Total Knee Arthroplasty Patient
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Discharge to a sub-acute rehabilitation after arthroplasty surgery is discouraged after due to the pandemic. The protocol is being revised to remove this arm of the study.
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-0907
Record Dates: First submitted 2020-11-23; First posted 2020-12-07 (Actual); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Total Knee Replacement
Keywords: Total Knee Replacement; Postoperative Rehabilitation; Total Knee Arthroplasty

STUDY DESIGN:
Intervention Model Description: DJO X4 Brace with Motion Intelligence Platform: Home discharge. Patients randomized to this group will be provided with the X4 brace and trained on the use of Motion Intelligence platform.
  Control group: Home discharge. Patients randomized to this group will serve as the control group. There will be no changes to the standard of care recovery for a TKA patient.
  DJO X4 Brace with Motion Intelligence Platform: Discharge to rehabilitation center. Patients randomized to this group will be provided with the X4 brace and trained on the use of Motion Intelligence platform.
  Cohort 4- Control group: Discharge to rehabilitation center. Patients randomized to this group will serve as the control group. There will be no changes to the standard of care recovery for a TKA patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- DJO X4 Brace with Motion Intelligence Platform: Home discharge (Experimental): Patients randomized to this group will be provided with the X4 brace and trained on the use of Motion Intelligence platform.
  Interventions: Device: DJO X4 brace with Motion Intelligence Platform
- Control group: Home discharge (No Intervention): Patients randomized to this group will serve as the control group. There will be no changes to the standard of care recovery for a TKA patient.
- DJO X4 Brace with Motion Intelligence Platform: Discharge to rehabilitation center (Experimental): Patients randomized to this group will be provided with the X4 brace and trained on the use of Motion Intelligence platform.
  Interventions: Device: DJO X4 brace with Motion Intelligence Platform
- Control group: Discharge to rehabilitation center (No Intervention): Patients randomized to this group will serve as the control group. There will be no changes to the standard of care recovery for a TKA patient.

INTERVENTIONS:
Device: DJO X4 brace with Motion Intelligence Platform — The X4 Knee brace with the Motion Intelligence platform uses both a bio-measurement equipment with an interactive application thereby providing the patient with immediate feedback on their exercise regime. The X4 Knee brace is a postoperative brace worn by a patient to monitor compliance to prescribed protocol based on the movement and function of the knee joint. The device also connects wirelessly to a companion mobile application, Motion Intelligence, and streams both real-time and collected data for review and record collection. Prescribed exercises are uploaded into the patient application, with a number of the exercises actively tracked by the Mi360 sensor housed in the X4 brace. Compliance can be tracked by the physician in real-time between postoperative visits and any medical staff on a separate dashboard.
  Arms: DJO X4 Brace with Motion Intelligence Platform: Discharge to rehabilitation center; DJO X4 Brace with Motion Intelligence Platform: Home discharge

SUMMARY:
This is a single center, investigator initiated clinical trial using a FDA approved, marketed brace called DJO X4. This phase 4, prospective, randomized clinical trial is being conducted to evaluate the use of the X4 knee brace with the Motion Intelligence platform in patients having unilateral TKA. The study is designed to determine if using a "virtual rehabilitation" device leads to enhanced recovery following TKA by improving patient objective and subjective outcome measures.

DETAILED DESCRIPTION:
This is a prospective, randomized clinical trial to evaluate the use of the X4 knee brace with the Motion Intelligence platform in patients having unilateral TKA. This brace is a FDA approved, marketed product being used as per the manufacturer's (DJO) marketed indications. This study is designed to determine if using a "virtual rehabilitation" device leads to enhanced recovery following total knee arthroplasty by improving patient objective and subjective outcome measures. These outcomes will be collected using a validated tool called the Knee Society Score (KSS). The KSS is a standard of care tool collected for all TKA patients pre-operatively and postoperatively at the 8 week visit.

Patients will be randomized to one to 4 cohorts:

DJO X4 Brace with Motion Intelligence Platform: Home discharge-Home. Patients randomized to this group will be provided with the X4 brace and trained on the use of Motion Intelligence platform.

Control group-Home discharge. Patients randomized to this group will serve as the control group. There will be no changes to the standard of care recovery for a TKA patient.

DJO X4 Brace with Motion Intelligence Platform: Discharge to rehabilitation center. Patients randomized to this group will be provided with the X4 brace and trained on the use of Motion Intelligence platform.

Cohort 4- Control group: Discharge to rehabilitation center. Patients randomized to this group will serve as the control group. There will be no changes to the standard of care recovery for a TKA patient.

The DJO X4 brace will be provided to the patient at no cost. Study visits, hospitalization, inpatient and outpatient rehabilitation costs are standard of care and will be the responsibility of the patient. There will be no payment for participation in this study.

All study patients will complete a daily "Daily Patient Log" starting the day after discharge from the hospital until postoperative day (POD) 56. This log will document the patient's location:

* Rehabilitation center or
* Home physical therapy or
* Physical therapy center
* Hospital (re-admission)
* Return to work (if applicable)

The study hypotheses is that the X4 brace with the Motion Intelligence platform will provide an enhanced, cost-effective postoperative recovery following total knee arthroplasty (TKA).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 or < 90
* Able to read and speak in English
* Patients having a unilateral total knee arthroplasty by Drs. Krauss or Segal
* Patients with a smart phone and internet able to access the Motion Intelligence Platform
* Patient is freely able to provide consent
* Patients willing to comply with the standard of care postoperative visit schedule (2 and 8 weeks)
* Agree to complete the KSS 2013 version preoperatively and at the 8 week postoperative visit
* Agree to complete the study required validated System Usability Scale at the 8 week postoperative visit

Exclusion Criteria

* Surgery covered by workman's compensation
* Physical impairments which in the opinion of the surgeon will effect or limit rehabilitation (e.g.: Multiple Sclerosis, Parkinson's disease)
* Limited mobility preoperatively requiring the use of a wheelchair
* Chronic opioid use prior to surgery
* Alcohol abuse
* Participation in another clinical trial
* Cognitive limitations which will interfere with the understanding of the Motion Intelligence platform
* Requirement for a knee immobilizer postoperatively

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene S Krauss, MD, Principal Investigator — Northwell Health System
Locations (1):
- Syosset Hospital, Syosset, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scuderi GR, Bourne RB, Noble PC, Benjamin JB, Lonner JH, Scott WN. The new Knee Society Knee Scoring System. Clin Orthop Relat Res. 2012 Jan;470(1):3-19. doi: 10.1007/s11999-011-2135-0. No abstract available. PMID 22045067

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group-Home Discharge.; Control Group-Discharge to Rehabilitation Center.: Patients randomized to this group will serve as the control group. There will be no changes to the standard of care recovery for a TKA patient.
Period: Overall Study
Arm/Group | DJO X4 Brace With Motion Intelligence Platform: Home Discharge | Control Group-Home Discharge. | DJO X4 Brace With Motion Intelligence Platform: Discharge to Rehabilitation Center | Control Group-Discharge to Rehabilitation Center.
Started | 8 | 8 | 0 | 0
Completed | 5 | 8 | 0 | 0
Not Completed | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated early. Only Cohorts 1 and 2 enrolled patients. There was no enrollment in Cohorts 3 or 4.
Groups:
- Cohort 1: Cohort 1- Study group-Home discharge. Patients randomized to this group will be provided with the X4 brace and trained on the use of Motion Intelligence platform.
  DJO X4 brace with Motion Intelligence Platform: The X4 Knee brace with the Motion Intelligence platform uses both a bio-measurement equipment with an interactive application thereby providing the patient with immediate feedback on their exercise regime. The X4 Knee brace is a postoperative brace worn by a patient to monitor compliance to prescribed protocol based on the movement and function of the knee joint. The device also connects wirelessly to a companion mobile application, Motion Intelligence, and streams both real-time and collected data for review and record collection. Prescribed exercises are uploaded into the patient application, with a number of the exercises actively tracked by the Mi360 sensor housed in the X4 brace. Compliance can be tracked by the physician in real-time between postoperative visits and any medical staff on a separate dashboard.
- Cohort 2: Cohort 2- Control group-Home discharge. Patients randomized to this group will serve as the control group. There will be no changes to the standard of care recovery for a TKA patient.
- Cohort 3: Cohort 3- Study group-Transfer to an inpatient rehabilitation center. Patients randomized to this group will be provided with the X4 brace and trained on the use of Motion Intelligence platform.
  DJO X4 brace with Motion Intelligence Platform: The X4 Knee brace with the Motion Intelligence platform uses both a bio-measurement equipment with an interactive application thereby providing the patient with immediate feedback on their exercise regime. The X4 Knee brace is a postoperative brace worn by a patient to monitor compliance to prescribed protocol based on the movement and function of the knee joint. The device also connects wirelessly to a companion mobile application, Motion Intelligence, and streams both real-time and collected data for review and record collection. Prescribed exercises are uploaded into the patient application, with a number of the exercises actively tracked by the Mi360 sensor housed in the X4 brace. Compliance can be tracked by the physician in real-time between postoperative visits and any medical staff on a separate dashboard.
- Cohort 4: Cohort 4- Control group-Transfer to an inpatient rehabilitation center. Patients randomized to this group will serve as the control group. There will be no changes to the standard of care recovery for a TKA patient.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 8 | 8 | 0 | 0 | 16
Age, Continuous [Mean (Full Range); unit: years] | 62 [52 to 72] | 61 [54 to 70] |  |  | 61.5 [52 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 |  |  | 6
  Male | 5 | 5 |  |  | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in the Calculated "Knee Society Score"
Description: Functional outcomes measured by the 2011 "Knee Society Score". The Functional Activities section consists of 4 sub-sections with a total score ranging from 0-100 points. The higher the numerical value the better the outcome. The sub-sections consist of: (1)Walking and Standing 0-30 points (2)Standard Activities 0-30 points (3)Advanced Activities 0-25 points (4)Discretionary Knee Activities 0-15 points.
Time Frame: Preoperatively and 8 weeks postoperatively
Population: The study was terminated early. In Cohort 1 only 3 patients completed the postoperative Knee Society Score. In Cohort 2 only 4 patients completed the postoperative Knee Society Score. Cohort 3 and 4 enrolled no patients.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 4
score on a scale | 59.7 [50 to 78] | 60.5 [34 to 83]

ADVERSE EVENTS:
Time Frame: Data was collected for 2 months postoperatively.
Description: 16 patients were enrolled in the study when the study was terminated. None of these patients experienced any device related adverse events.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT04655703/Prot_SAP_000.pdf